CLINICAL TRIAL: NCT04379986
Title: Remote Blood Pressure Monitoring With the Wearable SENBIOSYS Photoplethysmographic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stéphane Cook, Prof (Other)
Responsible Party: Sponsor-Investigator, Stéphane Cook, Prof, Clinical Professor, University of Freiburg
Organization: University of Freiburg (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SENBIOSYS trial
Record Dates: First submitted 2020-04-22; First posted 2020-05-08 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2020-05

CONDITIONS: Blood Pressure
Keywords: blood pressure; remote monitoring; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized measures in the cardiac catheterization laborator (Experimental): Immediately after coronary angiography, intra-arterial BP waveforms will be recorded using a fluid-filled catheter via right femoral or radial access. The catheter will be flushed before any waveform recordings is made. At first, the catheter will be positioned in the aorta for 3 minutes of stable BP waveforms recording. Intracoronary nitroglycerin will be administered at a dose of 300 µg, newly preceding 3 minute of recording. At the end of the coronary angiography, additional 3 minutes of recording will be performed in the aorta.
  Interventions: Device: Senbiosys
- Standardized measures in the intensive care unit (Experimental): Invasive BP monitoring is a commonly used technique in the ICU and is used to guide many intensive care unit therapies. Enrolled patients must have had an arterial catheter in place at the time of inclusion to the study. Arterial catheterization will be performed by the intensive care team according to current medical guidelines. No arterial catheters were placed for the sole purpose of this study. The Senbiosys device will be placed on the opposite arm of the arterial catheter for simultaneous measurements.
  Interventions: Device: Senbiosys

INTERVENTIONS:
Device: Senbiosys — The patients will undergo blood pressure estimation as per clinical routine and will simultaneously wear the device.

SUMMARY:
During the last couple of years, a growing number of wearable devices evolved to provide accurate, cheap and non-invasive monitoring of vitals parameters.This connected care technology could be helpful for treatment and care during a pandemic such as COVID-19. The use of these non-invasive remote monitoring devices can help health care providers to assess patient's vital signs and symptom progression, reducing reducing patient and healthcare provider contact and exposure to COVID-19 during this pandemic.

DETAILED DESCRIPTION:
Several cuff-less blood pressure monitoring devices have emerged in patient care using photoplethysmography. PPG utilizes an infrared or visible light to measure peripheral volumetric variations of blood circulation and its waveform has been proven to have a good correlation with BP waveform.Nonetheless, the accuracy of these instruments is of fundamental importance.

Several validation procedures for assessing the precision of BP monitoring devices have been developed, including protocols by the Association for the Advancement of Medical Instrumentation, International Organization for Standardization and European Society of Hypertension. Adherence to these guidelines are essential to ensure the effectiveness of BP measurement of the wearable devices.

Therefore, the investigators propose to test wearable low-noise, low-power SENBIOSYS photoplethysmography signals for estimation of BP.

ELIGIBILITY:
Participants fulfilling the following inclusion criteria are eligible for the study:

* Age ≥ 18 years
* Patients referred for coronarography
* Patient in the intensive care unit requiring invasive blood pressure monitoring and with an arterial catheter in place at the time of inclusion to the study

The presence of any of the following exclusion criteria will lead to exclusion of the participant:

* Unable or unwilling to provide written informed consent
* Coronarography in patients with myocardial infarction
* Patient with suspected or certified COVID-infection
* Patients with atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of non-invasive BP monitors: blood pressure | 10 to 15 minutes per patient (once)
  The primary outcome is the assessment of mean bias (± 95% CI or precision of bias) for systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean blood pressure (MBP) between invasive and non-invasive BP measurements. The standard deviation of the bias (±95% limits of agreement), will be assessed for SBP, DBP, and MBP measurements.

SECONDARY OUTCOMES:
Percentage of signal with artefact, | 10 to 15 minutes per patient (once)
  Secondary outcomes include reliability index (Qualification Index QI) for blood pressure epochs and count of qualified epochs.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Cook, MD, Study Chair — University of Freiburg
Locations (1):
- University and hospital Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Watanabe N, Bando YK, Kawachi T, Yamakita H, Futatsuyama K, Honda Y, Yasui H, Nishimura K, Kamihara T, Okumura T, Ishii H, Kondo T, Murohara T. Development and Validation of a Novel Cuff-Less Blood Pressure Monitoring Device. JACC Basic Transl Sci. 2017 Dec 25;2(6):631-642. doi: 10.1016/j.jacbts.2017.07.015. eCollection 2017 Dec. PMID 30062178
- [Result] Smolle KH, Schmid M, Prettenthaler H, Weger C. The Accuracy of the CNAP(R) Device Compared with Invasive Radial Artery Measurements for Providing Continuous Noninvasive Arterial Blood Pressure Readings at a Medical Intensive Care Unit: A Method-Comparison Study. Anesth Analg. 2015 Dec;121(6):1508-16. doi: 10.1213/ANE.0000000000000965. PMID 26496367
- [Result] Martinez G, Howard N, Abbott D, Lim K, Ward R, Elgendi M. Can Photoplethysmography Replace Arterial Blood Pressure in the Assessment of Blood Pressure? J Clin Med. 2018 Sep 30;7(10):316. doi: 10.3390/jcm7100316. PMID 30274376
- [Derived] Schukraft S, Boukhayma A, Cook S, Caizzone A. Remote Blood Pressure Monitoring With a Wearable Photoplethysmographic Device (Senbiosys): Protocol for a Single-Center Prospective Clinical Trial. JMIR Res Protoc. 2021 Oct 7;10(10):e30051. doi: 10.2196/30051. PMID 34617912